CLINICAL TRIAL: NCT04065100
Title: Sebum Measurement in Newborn to Detect Hyperexposure to Androgens
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Homerton University Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 120853
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Intervention Model Description: pregnant women with and without PCOS will be recruited in mid pregnancy. the newborn will be examined for sebum production and the two groups compared with each other and with and maternal testosterone levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Maternal PCOS
  Interventions: Diagnostic Test: Sebum test
- Comaprator (Active Comparator): Non-PCOS pregnant women
  Interventions: Diagnostic Test: Sebum test

INTERVENTIONS:
Diagnostic Test: Sebum test — Measuring sebum in newborn
  Other Names: Sebum measurements

SUMMARY:
The source of PCOS is unknown. Our hypothesis is that over exposure to testosterone of the foetus in utero alters the expression of genes thought to be involved in the cause of PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) affecting 10-15% of the female population causes excess hair, acne, irregular/absent ovulation, infertility and is associated with hypertension, diabetes, heart attacks and stroke in later life.

The economic care-related burden of the syndrome is estimated at $4.36 billion/year in the USA. The root cause is unknown and although mostly familial, the offending genes are unknown. We believe that excess testosterone, to which the foetus is exposed during its life in the womb, causes development of PCOS in adult life. If a mother with PCOS exposes her foetus to high testosterone levels compared to one with no PCOS, this would be the first step in proving the developmental hypothesis for PCOS, opening the door to methods to prevent the appearance of the distressing symptoms of PCOS in adult life.

With no access to the foetal environment, we have used the surrogate measure of sebum on the skin of the newborn, 99% influenced by testosterone. Our pilot study (Homburg et al, 2017) used absorbent paper to measure sebum excretion in PCOS and controls within 24 hours and 1-24 weeks after birth in mother and baby. Higher sebum production in female babies of PCOS mothers strongly supported our hypothesis.

The present proposal utilizes a 30-second, non-invasive, quantitative measurement of sebum (Sebumeter®) in the newborn from PCOS mothers and controls, within 24 hours of birth. We will correlate results with other features in both female and male newborn that may suggest hyper-exposure to testosterone and with maternal testosterone levels in the blood. If confirming the findings of our pilot study in line with the developmental theory of PCOS, this could be used within 24 hours of birth to predict development of PCOS in adult life, induce measures to prevent the symptoms of PCOS and reduce the enormous health burden on patients and economies

ELIGIBILITY:
Inclusion Criteria:

Women (with and without a diagnosis of polycystic ovarian syndrome) aged 18-40 with an uncomplicated singleton pregnancy, who deliver a baby at term (37 weeks gestation or longer). Women in the PCOS cohort will be defined by the ESHRE/ASRM Rotterdam criteria. Women with no signs of PCOS who deliver a term baby will serve as the control group.

Exclusion Criteria:

Patients who decline consent

Ages: 30 Minutes to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Sebum secretion | 30 seconds
  Do term babies of mothers with PCOS have significantly increased sebum output in the neonatal period compared with those from mothers without PCOS

SECONDARY OUTCOMES:
Maternal testosterone levels | 1 minute
  The correlation between the maternal blood levels of androgens during pregnancy and the quantity of sebum produced by the newborn?
Ano-genital distance and finger length in the newborn | 15 minute
  Correlation of the level of sebum production in the neonate with other measures (ano-genital distance, finger lengths) of androgen exposure of the foetus during pregnancy?

CONTACTS AND LOCATIONS:
Overall Officials: Roy Homburg, Study Director — Homerton University Hospital NHS Foundation Trust
Locations (1):
- Homerton Fertility Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
May share after publication.